CLINICAL TRIAL: NCT05737472
Title: A Proof-of-concept Randomized Control Trial on the Role of Higher Protein Quantity and Quality-ready-to-use Therapeutic Food in Improving Linear Growth Among 6-23-month-old Children With Severe Wasting
Brief Title: High-protein Quantity and Quality RUTF in Improving Linear Growth Among Children With Severe Wasting
Acronym: Protein+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Ministry of Health, Malawi (Other Government); Schlumberger Foundation (Unknown); Nutriset (Industry); Friends of Sick Children, Malawi (Unknown)
Responsible Party: Principal Investigator, Robert Bandsma, Associate Professor, Staff Gastroenterologist, Principal Investigator, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1000079230
Record Dates: First submitted 2022-12-21; First posted 2023-02-21 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Severe Wasting; Severe Acute Malnutrition
Keywords: Child health; Ready-to-use therapeutic food; Severe acute malnutrition; RUTF; SAM; Wasting; Outpatient Therapeutic Programme; OTP
MeSH Terms: conditions — Cachexia; Severe Acute Malnutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patients, investigators, care providers, and data analysts will be blinded from the treatment allocation until data analysis is complete, thus quadruple blinding. The two RUTFs will be packaged in identical 92g sachets. The RUTFs will be as similar as possible in colour, texture, and smell. The two packages/sachets of the two types of RUTF will differ by colour, and the number code will be either grey-88 or purple-99 (the colour code will be unique to each RUTF type). An independent statistician will perform the colour allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard RUTF (Active Comparator): The standard RUTF dose is according to weight as per the WHO 2013 guideline, thus 150-220Kcal/kg/day. A child will receive a weekly ration for 8 consecutive weeks from enrolment.
  Interventions: Dietary Supplement: Standard RUTF
- High-protein RUTF (Experimental): The high-protein RUTF dose is according to weight as per the WHO 2013 guideline, thus 150-220Kcal/kg/day. A child will receive a weekly ration for 8 consecutive weeks from enrolment.
  Interventions: Dietary Supplement: High-protein RUTF

INTERVENTIONS:
Dietary Supplement: High-protein RUTF — The high-protein RUTF is isocaloric to the standard RUTF. To have a higher protein quantity and quality, the recipe has greater proportions of milk powder plus whey protein and vegetable oil. A total of 15% of energy is from protein. The protein quality score, digestible indispensable amino acid score (DIAAS )of the high protein, RUTF is 1.18 which is equivalent to a Protein Digestibility Corrected Amino Acid Score (PDCAAS) of 1.19
  Arms: High-protein RUTF
Dietary Supplement: Standard RUTF — The standard RUTF was manufactured according to WHO recommendations, with at least 50% of protein-sourced dairy, mainly skim milk. A total of 10% of energy is from protein. The protein quality score, digestible indispensable amino acid score (DIAAS) of the standard RUTF is 0.76, which is equivalent to a Protein Digestibility Corrected Amino Acid Score (PDCAAS) of 0.86.
  Arms: Standard RUTF

SUMMARY:
This is a proof-of-concept trial that aims to compare the efficacy of an 8-week treatment with higher-protein-Ready-to-Use Therapeutic Foods (RUTF) with standard RUTF in improving levels of markers of growths, height, nutritional recovery, and lean mass deposition among children with severe wasting. The study will also assess the safety and acceptability of the high-protein RUTF in comparison to the standard RUTF. The study will be conducted at four outpatient therapeutic programs in the Blantyre district of Malawi.

DETAILED DESCRIPTION:
RUTF has successfully promoted recovery from severe wasting and widened treatment coverage. However, RUTF does not sufficiently promote linear growth, leaving many survivors of severe wasting at risk of persistent stunting. Stunting is associated with long-term effects like poor child development and an increased risk of non-communicable diseases in adults. High protein quantity and quality are known to stimulate linear growth; however, an RUTF with a higher protein quantity and quality than the standard RUTF has yet to be tested. The investigators hypothesize that the suboptimal linear growth in children surviving severe malnutrition can be improved by increasing the protein quantity and quality in the standard RUTF formulation. The investigators have designed a high protein quantity and quality RUTF that will be tested in a proof-of-concept quadruple-blind randomised controlled trial study design. The trial aims to compare the efficacy of higher-protein-RUTF and standard RUTF in improving markers of linear growth among 6-23 months old children with severe wasting.

Children aged 6-23 months newly enrolled in outpatient treatment programs for severe wasting and without medical complications are eligible. They will be assigned to either increased protein RUTF or standard RUTF for eight weeks.

The primary outcome is a change in insulin-like growth factor-1 (IGF- 1) after four weeks of treatment. IGF-1 is a hormone that is mechanistically linked with growth. Secondary outcomes include ponderal and linear growth changes from baseline measured at eight weeks and plasma amino acid profile at four weeks. Other secondary outcomes are the acceptability and safety of high protein RUTF compared to standard RUTF. These findings will help to determine the optimal protein composition of RUTF to promote linear growth when treating severe wasting in children.

ELIGIBILITY:
Inclusion Criteria:

* Infants 6-23 months of age with severe wasting at OTP admission according to the WHO criteria: WHZ below -3 or MUAC below 115mm.
* Parent or guardian is able and available to consent
* Children who are able to feed orally in the usual state of health
* The primary caregiver plans to stay in the study area during the duration of the study.

Exclusion Criteria:

* Children with medical complications as per the CMAM guidelines (lack of appetite, severe oedematous malnutrition, acute infections)
* mild and moderate nutritional oedema
* Children with a known terminal illness (e.g. cancer), cerebral palsy (CP), tuberculosis (TB,) HIV infected or exposed
* Children who had SAM in the last 8 weeks, i.e., SAM relapses in the last 8 weeks
* Children admitted to any NRU due to complicated SAM in the previous 4 weeks will also be excluded
* Children whose caregivers refuse to give consent or whose primary givers are not available to give consent
* Children who were previously enrolled in this trial or currently enrolled in this trial whose sibling has also been enrolled in the study
* Children with known intolerance or allergy to high protein diets will be excluded as well as known intolerance or allergy to milk/lactose

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-08-23 (Actual)

PRIMARY OUTCOMES:
Changes in plasma IGF-1 | 4 weeks
  To assess the efficacy of high-protein-RUTF with higher protein quality and quantity compared to standard RUTF in increasing circulating IGF- 1 in 6-23-month-old children with severe wasting.

SECONDARY OUTCOMES:
Changes in height for age z score | 8 weeks
  To assess the efficacy of high-protein-RUTF with higher protein quality and quantity compared to standard RUTF in improving change in height-for-age z score.
Changes in weight for age z score | 8 weeks
  To assess the efficacy of high-protein-RUTF with higher protein quality and quantity compared to standard RUTF in improving change in weight for age z score
Changes in weight for height z score | 8 weeks
  To assess the efficacy of high-protein-RUTF with higher protein quality and quantity compared to standard RUTF in improving change in weight for height z score
Changes in knee heel length | 8 weeks
  To assess the efficacy of high-protein-RUTF with higher protein quality and quantity compared to standard RUTF in improving change in knee heel length
Changes in plasma essential amino acid profile leucine, threonine and tryptophan | 4 weeks
  To assess the efficacy of high-protein-RUTF with higher protein quality and quantity compared to standard RUTF in improving plasma essential amino acids: leucine, threonine and tryptophan
Changes in IGFBP3 | 4 weeks
  To assess the efficacy of high-protein-RUTF with higher protein quality and quantity compared to standard RUTF in increasing IGFFBP3
Changes in fat free mass accretion | 8 weeks
  • To assess the efficacy of high-protein-RUTF with higher protein quality and quantity compared to standard RUTF in improving fat free mass accretions (kg/m2) using bioelectrical impedance and skinfold thickness
Changes in fat mass accretion | 8 weeks
  • To assess the efficacy of high-protein-RUTF with higher protein quality and quantity compared to standard RUTF in improving fat mass accretion (kg/m2) using bio-electrical impedance assessment and skinfold thickness
Acceptability of high-protein RUTF | 4
  • To assess acceptability of the high protein RUTF formulation compared to standard RUTF among children with severe wasting using an adaptation of action against hunger RUTF apettite test
Acceptability of high-protein RUTF | 4
  • To assess acceptability of the high protein RUTF formulation compared to standard RUTF among children with severe wasting by observing RUTF intake at participant homes for 5 hours at a single time point
Compliance of high-protein RUTF | 4
  • To assess compliance of the high protein RUTF formulation compared to standard RUTF among children with severe wasting by conducting in-depth interviews with the caregivers
Safety of the high protein RUTF formulation:adverse events | 8 weeks
  To assess the safety of high-protein-RUTF compared to standard RUTF by recording adverse events (defined as any untoward event including morbidity reported by the participant or detected by the investigator)
Safety of the high protein RUTF formulation: severe adverse events | 8 weeks
  To assess the safety of high-protein-RUTF compared to standard RUTF by recording adverse events (defined as any life threatening event reported by the participant or detected by the investigator)

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Potani, PhD(c), Principal Investigator — The Hospital for Sick Children
Locations (1):
- Ndirande, Mbayani, Bangwe, Limbe and Bangwe health centres, Blantyre, Malawi

IPD SHARING:
Plan to Share IPD: No
De-identified data may be made available after publication of the results in line with the study's sponsor's procedures for release.

REFERENCES:
- [Background] Potani I, Spiegel-Feld C, Brixi G, Bendabenda J, Siegfried N, Bandsma RHJ, Briend A, Daniel AI. Ready-to-Use Therapeutic Food (RUTF) Containing Low or No Dairy Compared to Standard RUTF for Children with Severe Acute Malnutrition: A Systematic Review and Meta-Analysis. Adv Nutr. 2021 Oct 1;12(5):1930-1943. doi: 10.1093/advances/nmab027. PMID 33838044
- [Background] Shivakumar N, Jackson AA, Courtney-Martin G, Elango R, Ghosh S, Hodgkinson S, Xipsiti M, Lee WTK, Kurpad AV, Tome D. Protein Quality Assessment of Follow-up Formula for Young Children and Ready-to-Use Therapeutic Foods: Recommendations by the FAO Expert Working Group in 2017. J Nutr. 2020 Feb 1;150(2):195-201. doi: 10.1093/jn/nxz250. PMID 31724705
- [Derived] Potani I, Daniel AI, Briend A, Courtney-Martin G, Berkley JA, Voskuijl W, Vresk L, Bourdon C, Kathumba S, Mbale E, Bandsma RHJ. A protocol for a proof-of-concept randomized control trial testing increased protein quantity and quality in ready-to-use therapeutic food in improving linear growth among 6-23-month-old children with severe wasting in Malawi. PLoS One. 2023 Aug 24;18(8):e0287680. doi: 10.1371/journal.pone.0287680. eCollection 2023. PMID 37619218